CLINICAL TRIAL: NCT02670070
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics, Safety, and Tolerability of the Combination of Gemigliptin/Rosuvastatin 50/20 mg in Comparison to Each Component Gemigliptin 50 mg and Rosuvastatin 20 mg Administered in Healthy Male Volunteers
Brief Title: BE Study of the Combinations of Gemigliptin 50mg and Rosuvastatin 20mg in Comparison to Each Component Administered Alone
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-GSCL003
Record Dates: First submitted 2015-12-22; First posted 2016-02-01 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coadministration of G+R (Active Comparator): Coadministration of gemigliptin 50mg and rosuvastatin 20mg
  Interventions: Drug: gemigliptin 50mg, rosuvastatin 20mg
- Combination G/R (Experimental): Combination of gemigliptin 50mg / rosuvastatin 20mg
  Interventions: Drug: gemigliptin 50mg, rosuvastatin 20mg

INTERVENTIONS:
Drug: gemigliptin 50mg, rosuvastatin 20mg — gemigliptin/rosuvastatin 50/20mg
  Other Names: Zemiglo, Cresto

SUMMARY:
This study is to evaluate the safety/tolerability and pharmacokinetics of the combinations of gemigliptin 50mg and rosuvastatin 20mg in comparison to each component administered alone in healthy male volunteers.

DETAILED DESCRIPTION:
This study is to evaluate the safety/tolerability and pharmacokinetics(AUC and Cmax) of the combinations of gemigliptin 50mg and rosuvastatin 20mg in comparison to each component administered alone in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 45, healthy male subjects(at screening)
* BMI between 18.0 - 27.0
* FPG 70-125mg/dL glucose level(at screening)
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology,immunology,pulmonary,endocrine,hematooncology,cardiology,mental disorder.)
* Subject who had GI tract disease or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
* Subject who had drug hypersensitivity reaction.(Aspirin, antibiotics)
* Subject who already participated in other trials in 2months
* Subject who had whole blood donation in 2 months, or component blood donation in 1 month or transfusion in 1 month currently.
* Heavy smokers.(>10 cigarettes per day)

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
AUClast, Cmax | up to 72h post-dose
  To evaluate AUClast/Cmax of gemigliptin and rosuvastatin

SECONDARY OUTCOMES:
AUCinf | up to 72h post-dose
  To evaluate AUCinf of gemigliptin, LC15-0636 of gemigliptin metabolite and rosuvastatin
Tmax | up to 72h post-dose
  To evaluate Tmax of gemigliptin, LC15-0636 of gemigliptin metabolite and rosuvastatin
t1/2 | up to 72h post-dose
  To evaluate t1/2 of gemigliptin, LC15-0636 of gemigliptin metabolite and rosuvastatin
CL/F | up to 72h post-dose
  To evaluate CL/F of gemigliptin, LC15-0636 of gemigliptin metabolite and rosuvastatin
metabolic ratio | up to 72h post-dose
  To evaluate metabolic ratio of gemigliptin, LC15-0636 of gemigliptin metabolite
AUEC | up to 72h post-dose
  This parameter is been used to measure pharmarcodynamic characters of gemigliptin, the supression rate of DPP4 activity.
Emax | up to 72h post-dose
  This parameter is been used to measure pharmarcodynamic characters of gemigliptin, the supression rate of DPP4 activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No